CLINICAL TRIAL: NCT05584085
Title: The Effects of Acceptance-based Diabetes Education on Diabetes Distress and Glycaemic Control in Adults With Type 2 Diabetes: A Randomised Controlled Trial.
Brief Title: ACT-DE for Diabetes Distress and HbA1c in Adults With Type 2 Diabetes
Acronym: ACT-DE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anna Ngan, Principle Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACT-DE for DD and HbA1c
Record Dates: First submitted 2022-10-05; First posted 2022-10-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acceptance and Commitment Therapy; Diabetes Education; Diabetes Distress; HbA1c; Psychological Flexibility; Diabetes Self-management; Diabetes Management Self-efficacy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated (1:1 ratio) to either the intervention group that receive 1 6-week ACT-DE programme, while participants in the control group receive one session of diabetes education.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor who is responsible for collecting outcome data and data entry has no idea about the group allocation or participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and commitment therapy integrated in diabetes education (ACT-DE) (Experimental): The proposed intervention is a six-week acceptance-based diabetes education programme (ACT-DE) comprising acceptance and commitment therapy and diabetes education.
  Session 1: Diabetes education and introduction of ACT-DE programme Session 2: Mindfulness cultivation Session 3: Value clarification Session 4: Integrating ACT into diabetes self-management Session 5: Booster session Session length: 120 minutes Group-based (6-8 participants) and face-to-face mode of delivery
  Interventions: Behavioral: ACT-DE
- Diabetes education (Placebo Comparator): One session of diabetes education, group-based (6-8 participants) and 120 minutes via face-to-face delivery.
  Interventions: Behavioral: ACT-DE

INTERVENTIONS:
Behavioral: ACT-DE — Acceptance and Commitment Therapy is a third-wave psychological therapy to cultivate participants' acceptance attitude to diabetes and motivate them for a value-driven persistent diabetes self-management, directed by six psychological processes in the ACT hexagonal model, including acceptance, cognitive defusion, the present moment, self-as-context, value clarification and committed action.

SUMMARY:
This study will evaluate the effectiveness of a structured acceptance-based diabetes education programme for adults with type 2 diabetes compared with those who received diabetes education. The programme mainly comprises acceptance and commitment therapy (ACT) as a psychological component and a diabetes education (DE) component. The short form of the programme is named 'ACT-DE'. This programme aims to decrease the diabetes distress level in participants with type 2 diabetes and improve their blood glucose level. The objectives are:

1. To develop an ACT-based intervention protocol as a guide for promoting healthy coping in people with type 2 diabetes who are psychologically distressed.
2. To examine the effects of 'ACT-DE' on diabetes distress and HbA1c (primary outcomes) over a three-month follow-up, when compared with diabetes education only.
3. To examine the effects of 'ACT-DE' on diabetes self-management behaviours, self-efficacy in diabetes care, and psychological flexibility (secondary outcomes) over the three-month follow-up, when compared with diabetes education; and
4. To identify the relationships between psychological flexibility and diabetes self-efficacy, diabetes self-management behaviour and HbA1c among the study participants

DETAILED DESCRIPTION:
Diabetes distress is an aversive feeling and emotional disturbance specific to diabetes, including the burden of daily self-care, worry and guilty feelings, and low satisfaction level with health care professionals. Around 36% of people with type 2 diabetes worldwide suffered from diabetes distress, which is associated with poor self-care performance, low self-efficacy in diabetes management and higher blood glucose levels. Acceptance and commitment therapy, one of the mindfulness and acceptance-based interventions, integrated with diabetes education are found to be potentially effective interventions for reducing diabetes distress.

A pilot study has been conducted earlier (NCT05563987) and showed that a six-week ACT-DE programme (5 sessions) was preliminary effective compared to attending only one session of diabetes education. It was also a feasible and acceptable intervention.

In this main study, a convenience sampling method will be adopted from three out-patient clinics of public hospitals in Hong Kong. A total of 176 eligible participants will be randomly allocated into the intervention (N=88) and the control group (N=88). Participants in the intervention group will receive 6-week ACT-DE programme (5 sessions) composing acceptance and commitment therapy and diabetes education. Each session last for 120 minutes in a group of 8-10 participants. Participants in the control group will receive one session of diabetes education.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults Hong Kong Chinese residents,
* aged 18-64,
* diagnosed with type 2 diabetes for over one year;
* at least moderate level of diabetes distress as measured with the Chinese
* Diabetes Distress Scale (CDDS-15; mean score >2 per item);
* having suboptimal blood glucose control as shown by HbA1c level of ≥ 7% in the laboratory results within the past six months;
* able to communicate in Cantonese and give written consent

Exclusion Criteria:

* history of a clinically diagnosed mental illness such as depression and anxiety disorder, and/or an acute/severe medical disease;
* noticeable cognitive impairment(s) as indicated by the total score (<6 of 10) of the Abbreviated Mental Test;
* recently received/receiving any psychological therapy such as mindfulness or acceptance-based therapy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Diabetes Distress Scale at 3 months post intervention | Baseline (T0), immediate post-intervention (T1) and 3-month post-intervention (T2)
  Diabetes distress will be measured by the Chinese 15-item Diabetes Distress Scale (CDDS-15). It consists of 15 items.
  rated on a six-point Likert scale from 1 = 'not a problem' to 6 = 'a serious problem'. A mean item score of 2-2.9 and
  ≥3.0 indicates moderate and severe distress, respectively.
Change from baseline HbA1c at 3 months post-intervention | Baseline (T0), and 3-month post-intervention (T2)
  Blood glucose level of participants will be evaluated with an HbA1c level, which measures the average blood glucose level during the past three months. An HbA1c level over 7% is considered suboptimal glycaemic control, indicating a high risk of diabetes complications.2 HbA1c values obtained every 3-4 months will be collected from the patient electronic information system.

SECONDARY OUTCOMES:
Diabetes self-management behaviours | Baseline (T0), immediate post-intervention (T1) and 3-month post-intervention (T2)
  was measured by the Chinese version of diabetes self-management activities (C-SDSCA). It has 11 items rated on an eight-point Likert scale from 0 to 7, with higher scores indicating more attention to self-management activities.
Diabetes management self-efficacy | Baseline (T0), immediate post-intervention (T1) and 3-month post-intervention (T2)
  was measured by the Chinese version of Diabetes Management Self-Efficacy Scale (C-DMSES). The C-DMSES contains 20 items rated on an 11#point Likert scale, in which zero indicates not at all confident, and 10 indicates very confident.
Psychological flexibility | Baseline (T0), immediate post-intervention (T1) and 3-month post-intervention (T2)
  was measured by the Chinese version of the Acceptance and Action Questionnaire (AAQ-II Chinese). It contains seven items rated on a seven-point, agreement-based response scale from 1 = 'never true' to 7 = 'always true'. The
  - Page 3 of 5 - AAQ-II will be scored by summing all item responses, with higher scale scores indicating a greater psychological inflexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- The Nethersole School of Nursing, Hong Kong, Hong Kong Island, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided